CLINICAL TRIAL: NCT03120338
Title: eHealth Services for Child and Adolescent Psychiatry (eCAP): A Trial of the DAWBA as a Rapid Online Assessment Tool
Brief Title: DAWBA as a Rapid Online Assessment Tool
Acronym: eCAP:DAWBA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aberdeen (Other)
Collaborators: NHS Highland (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 17/NS/0002
Record Dates: First submitted 2017-04-10; First posted 2017-04-19 (Actual); Last update posted 2021-02-23 (Actual); Status verified 2021-02

CONDITIONS: Mental Health Services
Keywords: Child and Adolescent; Randomised Controlled Trial; Paediatrics; DAWBA; eHealth Services

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Single Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The Development and Wellbeing Assessment (Experimental): The Development and Wellbeing Assessment (DAWBA: http://www.dawba.com/) is a computerised structured instrument for gathering diagnostic data from parents or guardians, teachers and young people themselves.
  The DAWBA will be administered in addition to care as usual.
  Interventions: Diagnostic Test: The Development and Wellbeing Assessment
- Care as Usual (No Intervention): Care as usual

INTERVENTIONS:
Diagnostic Test: The Development and Wellbeing Assessment — The Development and Wellbeing Assessment (DAWBA: http://www.dawba.com/) is a computerised structured instrument for gathering diagnostic data from parents or guardians, teachers and young people themselves.
  Other Names: DAWBA
  Arms: The Development and Wellbeing Assessment

SUMMARY:
The European Union is funding this randomised trial in Scotland as part of the larger eCAP project (http://www.interreg-npa.eu/projects/funded-projects/project/139/). The need for psychiatric services for children and adolescents is usually greater than the services available. As well as this, in many cases, there is confusion as to which service the child or young person should be referred to. The way children and young people arrive at Child and Adolescent Mental Health Services (CAMHS) may therefore be relatively inefficient and families could suffer as a result of this inefficiency.

The use of a computerised structured questionnaire such as the Development and Well-being Assessment (DAWBA) offers the opportunity for these difficulties to be addressed, for the avoidance of 'inappropriate referrals' and for more rational use of resources. It is usually administered online through a secure internet portal. At the end of the data collection, a computerised summary is generated from the data given by all the informants and a child/adolescent psychiatrist lists the likely diagnosis or diagnoses in a summary of the case and gives his view about the next steps. This is then made available to the referrer. This community-based study aims to establish whether using the DAWBA in this way helps children and young people with mental health problems. The main objectives are to improve their mental health, reduce waiting times, change referral practice, increase satisfaction in services and improve cost effectiveness. The principal outcome measure will be parent-rated Strengths and Difficulties Questionnaire (SDQ) score 6 months after randomisation. Secondary outcome measures will include teacher and child-rated SDQ at 6 months and waiting times to services. The investigators will also record service use data and family out -of -pocket costs. A random sample of young people, family and referrers will be interviewed to explore satisfaction with service.

DETAILED DESCRIPTION:
This project will involve 246 participants in each centre (123 intervention, 123 control). Assuming 20% loss to follow-up (i.e. 197 completing) this will give 80% power at 5% significance to detect a moderate effect size of 0.4 in each participating centre. If the investigators assume that the typical SDQ Total Difficulties Score six months after referral is 15 points (the boundary between 'borderline' and 'abnormal' scores), then this would correspond to a difference between the groups of around 2 points which is probably near the lower limit of clinically significant change.

Patient / parent name and telephone number will be supplied to the National Health Service (NHS) Highland research nurse after verbal agreement is given to the referring practitioner that the parent is happy to be contacted to gain formal consent to participate in the project. These details (name and telephone number) will be supplied to enable the research nurse to initially make contact with each participant.

The research nurse will then telephone the parent (contact will be made with the parent first or the young person if aged 16 or over and either the young person or their parent is unwilling for their parent to participate). If the parent agrees, the participant information sheet and consent form will be emailed or posted to the family. Informed consent to participation in the study will be obtained from parents or legal guardians and young people aged 16 & 17, and young people aged 11 to 15 years will be asked for assent. Consent/assent will be requested to cover:

* Participation in the project;
* Completion of simple questionnaires at baseline and six months;
* Provision of relevant contact details (parents, teachers, young people);
* allowing requests for qualitative interviews;
* giving researchers access to service use data. The consent form will explain that the project is designed to find out whether doing a detailed mental health assessment before specialist involvement improves the speed and efficiency of service delivery for families (see attached information sheets).

On receipt of the completed consent forms in the post, the NHS research nurse will assign a study number to the family and will contact the university statistics department (in Aberdeen) by email for group allocation. Participants will be assigned at random either to have a DAWBA administered (by parents in every case, by teachers when possible and by young people aged 11 or over) plus usual care, or to receive usual care only.

If admitted into the project, participants' health records will be accessed by members of research team only to establish levels of service use before and following intervention. These data will be recorded as the number of contacts with a particular service e.g. General Practitioner (GP), school nurse, health visitor, Primary mental Health Worker (PMHW), social worker. No other details will be recorded.

All participants will then be asked to complete baseline measures including the Strengths and Difficulties Questionnaire (SDQ) and demographic (age, sex, family structure, socio-economic status, rurality/urban/city, and service use details. The investigators will ask for full postcodes to allow for Scottish Index of Multiple Deprivation (SIMD) rank to be ascertained. These baseline data will only be available to the study team (ideally collected via a secure web portal), and will not be seen by the local clinicians.

The DAWBA will be administered online whenever possible, but in cases where there are literacy problems or lack of internet connectivity, administration will be by telephone (the interview being conducted by one of the NHS research nurses). In the case of online completion, the NHS research nurse will pass on login details to parents, and ask them to pass these on to teachers and young people (where relevant). If the parents are not willing the NHS research nurse will do this. If the potential participant does not want information sent to anybody else, then the information will not be sent. The potential participant's wishes will be respected.

Once all assessments are completed, the NHS research nurse will alert the local DAWBA rater. DAWBA ratings will be done by a local psychiatrist familiar with diagnostic classification and local services. In exceptional circumstances (e.g., no psychiatrist available due to illness) the Chief Investigator (Phil Wilson) is authorised to rate DAWBAs. (As the online system is anonymised, this will not jeopardise his blindness to randomisation.) The summarised DAWBA data and the full report will be shared with the referring clinician. The referrer will make their own decision about how to handle communication about the DAWBA data with families, referrers and specialist services. Other data, including the SDQ, will be held securely and kept confidential by the research team as below.

Any data collected will be treated confidentially and will be reported anonymously. Any data collected will be adequate, relevant and not excessive to the purpose of the research study proposed.

All data will be retained according to the University of Aberdeen's retention policy.

The NHS Highland General Practitioners have full access to patient records as a matter of routine, the research nurses will have access to patient / parent or teacher name / telephone number. These NHS staff are familiar with handling data and operate under the umbrella of confidentiality legislation within the NHS.

Participant consent will be sought for the research team to have access to:

GP records, school nurse records, PMHW records, Health Visitor (in case of very young children) - to identify the number of times the participant has seen the referring professional or other mental health service providers during the six months post recruitment.

Normal clinical confidentiality will apply, specifically information will be stored in a locked filing cabinet or a password protected area of a shared drive within the University of Aberdeen network. Only direct members of the research team will have access to participant information and participants will be allocated a unique study number that does not contain identifiable information. Identifiable information will be stored separately from study information. Any identifiable data will be destroyed less than three months after the study has ended. All other data will be stored securely for 10 years. The Chief Investigator will act as custodian for all data. No personal identifiable information will be held on laptop computers.

All data will be archived at the University of Aberdeen according to University of Aberdeen policy.

Most data will be held within the secure server network of the University of Aberdeen. It is impossible to access server drives without a valid staff username and password, and all files will be held within a password protected area accessible only to members of the study team. Any paper based data (such as a contact list for participants) will be held in a locked filing cabinet at the Centre for Rural Health (University of Aberdeen) Data from the telephone interviews (undertaken by the study research nurse) will be stored centrally on a university held computer in accordance with University of Aberdeen data storage governance policies.

Data will be gathered in accordance to the terms of the Data Protection Act (1988).

Personal identifiers will not be stored with research data. Unique identification numbers will be used on separate contact information and research data files, which will be stored in separate, secure locations on the University of Aberdeen servers. The investigators will follow Data Protection Act and Caldicott guidelines in relation to use of patient information at all times.

Participants will complete the DAWBA online. To maximise confidentiality and keep potentially sensitive information safe, the DAWBA online system is anonymised - only the research group knows which child has which identifier. Additional security is provided by using a secure server with encryption.

Appropriate Child Protection training for the research nurses will be provided by NHS Highland, it will be a group session for everyone involved in the project. NHS Highland will keep the records of who has undertaken the training. There is also an independent contact for potential participants to go to throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be children, young people between the ages of 2 and 17 inclusive and their families at the first point at which contact with CAMHS is being considered by a health professional.

Exclusion Criteria:

* Lack of fluency in any of the languages available for DAWBA assessment which could be rated by members of the participating CAMHS services would be the only exclusion criterion.

Ages: 2 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 71 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Parent-rated Strengths and Difficulties Questionnaire | Six months post randomisation
  The Strengths and Difficulties Questionnaire (SDQ) is a brief behavioural screening questionnaire about 3-16 year olds. It exists in several versions to meet the needs of researchers, clinicians and educationalists.

SECONDARY OUTCOMES:
Child and teacher rated SDQ | Six months post randomisation
  The Strengths and Difficulties Questionnaire (SDQ) is a brief behavioural screening questionnaire about 3-16 year olds. It exists in several versions to meet the needs of researchers, clinicians and educationalists.
Waiting times | Six months post randomisation
  Waiting times to CAMHS first appointment (if any)
Service use costs | Six month post randomisation
  Estimated total service use costs across education, social care, all health (including CAMHS), and voluntary sector.
Onward referral | Six month post randomisation
  Whether or not referral to other agencies (including back to the referrer) took place

CONTACTS AND LOCATIONS:
Overall Officials: Phil Wilson, Principal Investigator — Centre for Rural Health, University of Aberdeen
Locations (1):
- Centre for Rural Health, Inverness, Highland, United Kingdom

IPD SHARING:
Plan to Share IPD: Yes